CLINICAL TRIAL: NCT02009878
Title: A Phase 1b, Multicenter, Pilot, Randomized, Double-blind Trial to Determine the Pharmacokinetics and Pharmacodynamics of Orally Administered Tolvaptan 3.75, 7.5, and 15 mg Tablets in Subjects With Syndrome of Inappropriate Antidiuretic Hormone Secretion
Brief Title: A PK Study of 3 Dosages of Tolvaptan in Patients With Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 156-12-203
Record Dates: First submitted 2013-12-09; First posted 2013-12-12 (Estimated); Results first posted 2016-05-16 (Estimated); Last update posted 2016-05-16 (Estimated); Status verified 2016-04

CONDITIONS: Syndrome of Inappropriate Antidiuretic Hormone Secretion (SIADH)
Keywords: SIADH
MeSH Terms: conditions — Inappropriate ADH Syndrome | interventions — Tolvaptan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- tolvaptan 3.75 mg (Other): tolvaptan 3.75 mg
  Interventions: Drug: tolvaptan
- tolvaptan 7.5 mg (Other): tolvaptan 7.5 mg
  Interventions: Drug: tolvaptan
- tolvaptan 15 mg (Other): tolvaptan 15 mg
  Interventions: Drug: tolvaptan

INTERVENTIONS:
Drug: tolvaptan — Subjects will receive a single dose of 3.75, 7.5 or 15 mg of tolvaptan on study Day 1
  Other Names: SAMSCA

SUMMARY:
This is a study to evaluate how the body handles and metabolizes (PK) the various doses of the drug Tolvaptan, and what the effect (PD) of the various doses of Tolvaptan are on the content of "salt" in blood and urine

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects greater than or equal to 18 years of age or the age of legal consent.
* Must have a BMI less than or equal to 32.0 kg/m2.
* Subjects must have a diagnosis of SIADH prior to randomization.
* Persistent euvolemic hyponatremia, evidenced by 3 serum sodium assessments of between 120 and 133 mmol/L, inclusive drawn locally as follows: one during the screening period, a second at check-in on Day -1, a third on Day 0 (12-24 hours prior to dosing), which will serve as the baseline value for efficacy endpoints
* Subjects with relatively intact renal function, ie, estimated glomerular filtration rate using the CKD-EPI formula of greater than or equal to 60 mL/min/1.73m2.
* Ability to provide written, informed consent prior to initiation of any trial related procedures, and ability, in the opinion of the PI, to comply with all the requirements of the trial.
* Sexually active males who are practicing a highly effective method of birth control during the trial and for 30 days after the last dose of trial medication or who will remain abstinent during the trial and for 30 days after the last dose, or sexually active females of childbearing potential who are practicing a highly effective method of birth control during the trial and for 30 days after the last dose of trial medication or who will remain abstinent during the trial and for 30 days after the last dose, or female subjects of nonchildbearing potential (surgically sterile or postmenopausal [1 year post menses]). If employing birth control, 1 of the following highly effective methods (failure rate <1%) must be used: vasectomy, tubal ligation, intrauterine device containing hormone (Mirena), combined oral contraceptive, hormone implants or hormone injections.

Exclusion Criteria:

* Daily use of diuretics within 14 days prior to screening assessments or randomization or the requirement for constant diuretic use for any reason.
* Clinically assessed hypovolemic state.
* Inability to respond to thirst.
* Subjects who cannot perceive thirst.
* Subjects with anuria.
* Urgent need to raise serum sodium acutely.
* Urinary outflow obstruction unless the subject is, or can be, catheterized during the trial.
* Severe hepatic impairment. Child-Pugh Class C (score of 10 or greater).
* Subjects who receive any medication given for the purpose of raising serum sodium while undergoing qualifying serum sodium assessments. Specifically: Hypertonic saline (including normal saline challenge) within 8 hours before each qualifying serum sodium screening assessment; Urea, lithium, demeclocycline, conivaptan, or tolvaptan within 4 days of each qualifying serum sodium screening assessment; Loop diuretics (eg. furosemide, bumetanide, torsemide) within 48 hours of each qualifying serum sodium screening assessment; Other treatment (including normal saline or oral sodium containing supplements) for the purpose of increasing serum sodium within 24 hours of each qualifying serum sodium screening assessment. Final determination will be made in consultation with the sponsor.
* Subjects with medication induced SIADH who have not been on stable medication for 3 months.
* CYP3A4 inhibitors taken within 5 elimination half-lives or within 96 hours of dosing, which ever time is longer. Final determination will be made in consultation with the sponsor.
* CYP3A4 inducers taken within 72 hours after 5 elimination half-lives (eg, rifampin, St. Johns Wort).
* Chemotherapy agents given in the previous 7 days prior to dosing or within 5 elimination half-lives of the agent; whichever is longer.
* Clinically significant abnormality in past medical history, or at the Screening physical examination, that in the investigator's or sponsor's opinion may place the subject at risk or interfere with outcome variables including absorption, distribution, metabolism, and excretion of drug. This includes, but is not limited to, history of or concurrent cardiac, hepatic, renal, neurologic, endocrine, GI, respiratory, hematologic, and immunologic disease.
* History of drug and/or alcohol abuse within 6 months prior to Screening.
* History of or current hepatitis or acquired immunodeficiency syndrome or carriers of HBsAg, anti-HCV, and/or HIV antibodies.
* History of any significant drug allergy.
* A positive alcohol test and/or drug screen for substance of abuse at Screening or upon Check-in to the clinical site.
* Subjects having taken an investigational drug within 30 days preceding trial entry.
* Any history of significant bleeding or hemorrhagic tendencies.
* A history of difficulty in donating blood.
* The donation of blood or plasma within 30 days prior to dosing.
* Consumption of alcohol and/or food and beverages containing methylxanthines, pomelo fruit, grapefruit, grapefruit juice, Seville oranges, or Seville orange juice within 72 hours prior to dosing.
* Exposure to any substances known to stimulate hepatic microsomal enzymes within 30 days prior to Screening (eg, occupational exposure to pesticides, organic solvents).
* Has Screening liver function values > 3 x ULN.
* Has primary polydipsia.
* Inability to take oral medications.
* Subjects who have supine blood pressure, after resting for greater than or equal to 3 minutes, higher than 140/90 mmHg or lower than 100/50 mmHg. The sponsor may allow exceptions if they are not deemed clinically significant.
* Subjects who have a supine pulse rate, after resting for greater than or equal to 3 minutes, outside the range of 40 to 90 bpm. The sponsor may allow exceptions significant.
* History of serious mental disorders that, in the opinion of the investigator, would exclude the subject from participating in this trial.
* Any subject who, in the opinion of the investigator, should not participate in the trial.
* Subjects who are pregnant or breastfeeding. A negative serum pregnancy test must be confirmed prior to randomization for all female subjects of childbearing potential.
* Subjects with Type 1 diabetes.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- Vseobecna fakultni nemocnice V Praze, Prague, Czechia
- Holstebro Regionhospital, Holstebro, Denmark
- Germany (5):
  - Medizinische Klinik im Klinikum Hannover, Hanover, Lower Saxony
  - Universitätsklinikum C.-G.-Carus, Dresden, Saxony
  - Evangelische Lungenklinik Berlin, Berlin
  - Universitaetsklinikum Koeln, Cologne
  - Universitaetsklinikum Schleswig-Holstein - Campus Luebeck, Lübeck
- Semmelweis Egyetem AOK, Budapest, Hungary
- Spain (2):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitario Clinico San Carlos, Madrid
- Sahlgrenska Universitetssjukhuset, Gothenburg, Sweden
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Royal Free Hospital, London
  - The Christie Hospital, Manchester

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted in 30 participants (29 received treatment) at 14 trial sites in 7 countries.
Pre-assignment Details: Participants with syndrome of inappropriate antidiuretic hormone secretion (SIADH) and a serum sodium concentration between 120 and 133 mmol/L were randomized to single doses of 3.75, 7.5, or 15 mg tolvaptan. Baseline pharmacodynamics (PD) was assessed for 24 hours predose. Pharmacokinetic (PK) and PD assessments were obtained 24 hours postdose.
Groups:
- Tolvaptan 3.75 mg: Participants had received a single dose of 3.75 mg oral tolvaptan.
- Tolvaptan 7.5 mg: Participants had received a single dose of 7.5 mg oral tolvaptan.
- Tolvaptan 15 mg: Participants had received a single dose of 15 mg oral tolvaptan.
Period: Overall Study
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Started | 10 | 11 | 9
Completed | 10 | 10 | 9
Not Completed | 0 | 1 | 0
Not completed — Participant Met Withdrawal Criteria | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: The baseline analysis population comprised of all participants who had taken one dose of the study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg | Total
Number analyzed (Participants) | 10 | 10 | 9 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.50 (8.66) | 70.20 (9.90) | 59.67 (15.43) | 66.34 (12.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 5 | 19
  Male | 4 | 2 | 4 | 10

OUTCOME MEASURES:

1. Primary Outcome: Maximal Increase From Baseline in Serum Sodium Concentration Following Tolvaptan Administration.
Description: Maximal increase in serum sodium is summarized below by tolvaptan dose. Blood samples for determination of plasma concentrations of tolvaptan were collected predose and at 1, 2, 3, 4, 6, 8, 12, 16, and 24 hours postdose on Day 1 or at Early Termination (ET).
Time Frame: Baseline to Day 2
Population: PD dataset comprised of all participants who had taken 1 dose of study medication and had all observed measurements.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Number analyzed (Participants) | 10 | 10 | 8
mmol/L | 3.6 (3.3) | 5.3 (2.5) | 7.9 (5.3)

2. Secondary Outcome: Cmax (Maximum (Peak) Plasma Concentration) for Tolvaptan in Plasma.
Description: Blood samples for determination of plasma concentrations of tolvaptan were collected predose and 1, 2, 3, 4, 8, 12, 16, and 24 hours postdose on Day 1 or at ET. PK parameters in participants with SIADH following tolvaptan administration for three different doses are presented below.
Time Frame: Baseline to Day 2
Population: PK parameter dataset comprised of all participants who had taken 1 dose of study medication and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Number analyzed (Participants) | 10 | 10 | 8
ng/mL | 37.7 (12.6) | 107 (48.9) | 157 (68.1)

3. Secondary Outcome: Tmax (Time to Maximum (Peak) Plasma Concentration) for Tolvaptan in Plasma
Description: as for outcome 2
Time Frame: Baseline to Day 2
Population: PK parameter dataset comprised of all participants who had taken 1 dose of study medication and had evaluable PK data.
Measure: Median (Full Range); unit: hours
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Number analyzed (Participants) | 10 | 10 | 8
hours | 1.50 [0.95 to 4.00] | 2.00 [1.00 to 4.00] | 2.00 [0.97 to 3.00]

4. Secondary Outcome: AUC Infinity (Area Under the Concentration-time Curve From Time Zero to Infinity) for Tolvaptan in Plasma
Description: Blood samples for determination of plasma concentrations of tolvaptan were collected predose and 1, 2, 3, 4, 8, 12, 16, and 24 hours postdose on Day 1 or at ET. If an indwelling catheter was utilized, saline flushes were used. PK parameters in participants with SIADH following tolvaptan administration for three different doses are presented below.
Time Frame: Baseline to Day 2
Population: PK parameter dataset comprised of all participants who had taken 1 dose of study medication and had evaluable PK data.
Measure: Mean (Standard Deviation); unit: ng·h/mL
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Number analyzed (Participants) | 10 | 10 | 8
ng·h/mL | 244 (90.7) | 655 (373) | 1000 (361)

5. Secondary Outcome: Change From Baseline in Serum Sodium Concentrations
Description: Samples were taken on Day 0 (baseline) at the corresponding Day 1 predose time and 12 hours postdose time; and on Day 1 at predose and at 2, 4, 6, 8, 12, and 24 hours postdose.
Time Frame: Baseline and Day 2
Population: PD dataset comprised of all participants who had taken 1 dose of study medication and had all observed measurements.
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Number analyzed (Participants) | 10 | 10 | 9
mmol/L
  (Day 0) 12 hour (N= 10, 9, 9) | -2.5 (1.3) | -2.3 (3.0) | -2.6 (2.2)
  (Day 1) 2 hour (N= 10, 10, 8) | -2.0 (4.4) | 2.4 (1.3) | 1.7 (1.8)
  (Day 1) 4 hour (N= 10, 10, 8) | -1.7 (4.7) | 3.5 (3.0) | 3.0 (2.3)
  (Day 1) 6 hour (N= 10, 10, 8) | -0.1 (4.7) | 3.1 (3.1) | 5.3 (4.2)
  (Day 1) 8 hour (N= 10, 10, 8) | 0.0 (4.8) | 3.2 (1.9) | 5.4 (4.6)
  (Day 1) 12 hour (N= 9, 10, 9) | -0.6 (4.5) | 3.6 (1.8) | 5.9 (4.7)
  (Day 1) 24 hour (N= 10, 10, 9) | 2.9 (3.8) | 4.6 (1.9) | 7.4 (4.8)

6. Primary Outcome: Time of Maximal Increase From Baseline in Serum Sodium Concentration Following Tolvaptan Administration.
Description: Time of maximal increase in serum sodium is summarized in the table below by tolvaptan dose. Samples were taken on Day 0 (baseline) at the corresponding Day 1 predose time and 12 hours postdose time; and on Day 1 at predose and at 2, 4, 6, 8, 12, and 24 hours postdose.
Time Frame: Baseline to Day 2
Population: PD dataset comprised of all participants who had taken 1 dose of study medication and had all observed measurements.
Measure: Median (Full Range); unit: hours
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Number analyzed (Participants) | 10 | 10 | 7
hours | 24.13 [2.03 to 24.25] | 6.38 [2.05 to 24.28] | 24.02 [6.25 to 24.30]

7. Secondary Outcome: Change From Baseline in Fluid Intake From 0-6 Hours, 0-12 Hours and 0-24 Hours
Description: Fluid intake was monitored on Day 0 (times relative to Day 1 dosing), and Day 1 at intervals of 0 to 6, 6 to 12, and 12 to 24 hours postdose. Fluid intake included fluid used for dosing (study medication and any concomitant medication); food items that included any significant amounts of water (e.g., Jello [including Gelatin and Jelly dessert] and soup) was added to the total fluid intake. Samples were taken on Day 0 (baseline) at the corresponding Day 1 predose time and 12 hours postdose time; and on Day 1 at predose and at 2, 4, 6, 8, 12, and 24 hours postdose.
Time Frame: Baseline and Day 2
Population: PD dataset comprised of all participants who had taken 1 dose of study medication and had all observed measurements.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Number analyzed (Participants) | 10 | 10 | 9
mL
  Day 1 (0 to 6 hour) | 97.5 (461.9) | -255.0 (257.3) | -103.0 (693.2)
  Day 1 (0 to 12 hour) | 210.0 (558.1) | -65.0 (566.4) | 118.8 (1019.6)
  Day 1 (0 to 24 hour) | 361.0 (647.0) | 129.0 (632.1) | 525.6 (1265.3)

8. Secondary Outcome: Change From Baseline in Fluid Balance (Fluid Intake Minus Urine Output) From 0-6 Hours, 0-12 Hours and 0-24 Hours.
Description: Fluid intake was monitored on Day 0 (times relative to Day 1 dosing), and Day 1 at intervals of 0 to 6, 6 to 12, and 12 to 24 hours postdose. Fluid intake included fluid used for dosing (study medication and any concomitant medication); food items that included any significant amounts of water (e.g., Jello [including Gelatin and Jelly dessert] and soup) was added to the total fluid intake. Urine was collected for baseline comparison on Day 0 for the 24 hour prior to Day 1 dosing at intervals of 0 to 2, 2 to 4, 4 to 6, 6 to 8, 8 to 12 hours, and 12 to 24 hours relative to the Day 1 dosing time. Fluid balance was determined as fluid intake minus urine output.
Time Frame: 2 days
Population: PD dataset comprised of all participants who had taken 1 dose of study medication and had all observed measurements.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Number analyzed (Participants) | 10 | 10 | 9
mL
  Day 1 (0 to 6 hour) | -403.7 (783.2) | -856.8 (528.1) | -1478.8 (958.6)
  Day 1 (0 to 12 hour) | -588.8 (1078.8) | -839.8 (553.7) | -1897.5 (1072.7)
  Day 1 (0 to 24 hour) | -278.3 (1171.7) | -537.8 (831.1) | -1700.6 (1301.3)

9. Secondary Outcome: Change From Baseline in Cumulative Urine Volume at 0-6 Hours, 0-12 Hours and 0-24 Hours.
Description: Urine was collected for baseline comparison on Day 0 for the 24 hour prior to Day 1 dosing at intervals of 0 to 2, 2 to 4, 4, to 6, 6, to 8, 8, to 12, and 12 to 24 hours relative to Day 1 dosing time. Urine was collected on Day 1 at intervals of 0 to 2,2 to 4, 4 to 6, 6 to 8, 8 to 12, and 12 to 24 hours postdose. For the start of the urine collection on Day 0, a window of 15 to 40 minutes prior to the assigned dosing time was acceptable, with the 0 to 24 hour collection period on Day 1 starting 24 hours after the start time on Day 0. Participants were asked to void immediately prior to the end of the collection interval. The volume of individual voids were measured and recorded prior to refrigerating. All voids in a collection interval were pooled at the end of the collection interval, at which time the volume was determined, recorded and an aliquot taken for osmolality, sodium, potassium, and creatinine assessments.
Time Frame: 2 days
Population: PD dataset comprised of all participants who had taken 1 dose of study medication and had all observed measurements.
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Number analyzed (Participants) | 10 | 10 | 9
mL
  Day 1 (0 to 6 hour) | 501.2 (584.4) | 601.8 (486.6) | 1375.6 (911.6)
  Day 1 (0 to 12 hour) | 798.8 (1024.4) | 774.8 (596.2) | 2016.3 (1668)
  Day 1 (0 to 24 hour) | 639.3 (1223.8) | 666.8 (732.3) | 2226.3 (2151.5)

ADVERSE EVENTS:
Time Frame: Adverse events were reported from the signing of the informed consent throughout the study and were followed for 7 (+2) days post last dose of study medication.
Groups:
- Tolvaptan 3.75 mg; Tolvaptan 7.5 mg; Tolvaptan 15 mg: Subjects will receive a single dose of 3.75, 7.5 or 15 mg of tolvaptan on study Day 1
Arm/Group | Tolvaptan 3.75 mg | Tolvaptan 7.5 mg | Tolvaptan 15 mg
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/10 | 1/9
Other Adverse Events (participants affected / at risk) | 0/10 | 1/10 | 3/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan 3.75 mg (N=10) | Tolvaptan 7.5 mg (N=10) | Tolvaptan 15 mg (N=9)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Tolvaptan 3.75 mg (N=10) | Tolvaptan 7.5 mg (N=10) | Tolvaptan 15 mg (N=9)
Dizziness (Nervous system disorders) | 0 | 1 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 1
Polyuria (Renal and urinary disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Center may publish study results but ≥ 60 days prior to any public presentation, a copy is sent to Sponsor for review and Center can delay publication for 60 days to permit Sponsor to protect its intellectual property rights or confidential information contained within the publication. The first publication is a joint publication, if Center is part of a multi-center study. Center is free to publish, if there is no multi-center publication within 18 months of completion/ termination of study.